CLINICAL TRIAL: NCT01861028
Title: Study Comparing Fit of the iTotal Versus Standard Total Knee Implants
Status: Terminated | Type: Observational
Why Stopped: Not enough patient volume to continue the study.
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-002
Record Dates: First submitted 2013-03-26; First posted 2013-05-23 (Estimated); Results first posted 2020-12-28 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis
Keywords: total knee replacement; total knee arthroplasty; patient-specific
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Phase I: A series of 50 consecutive primary iTotal patients will be compared to assess the fit of the tibial tray intra-operatively. These patients will have a series of tibial templates from Standard TKR implant sets trialed on the operative knee. Each template will be optimally sized and positioned based on the surgeon's judgment. Implant fit data (overhang and underhang) on the tibia for all templates will be taken from intra-operative measurements
- Phase II: The Phase I (50 consecutive primary iTotal patients) will also have implant fit data assessed for the femur. After final implantation is complete measurement will be assessed and recorded. A series of 25 primary knees that are scheduled for Standard TKR implants will then undergo the same measurements of the femur.

SUMMARY:
This study compares intraoperative fit of the patient-specific iTotal knee replacement to other standard knee replacement implants

DETAILED DESCRIPTION:
The study is designed as a single center, two arm analysis. The study will be completed in two phases, based on measurement type.

All additional data will be obtained from pre and post-operative subject surveys, operative and discharge records and radiographs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for a standard total knee replacement
* Patient who are scheduled for patient-specific total knee replacement (iTotal)
* Patient age > 18 years

Exclusion Criteria:

* Patients who do not receive a total knee replacement
* Unwilling or unable to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving either a standard total knee implant or an iTotal patient-specific total knee implant
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2013-02; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Martin, MD, Principal Investigator — JFK Medical Center
Locations (1):
- JFK Medical Center, Atlantis, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- iTotal CR TKR: A series of 44 consecutive primary iTotal patients will be compared to assess the fit of the tibial tray intra-operatively. These patients will have a series of tibial templates from Standard TKR implant sets trialed on the operative knee. Each template will be optimally sized and positioned based on the surgeon's judgment. Implant fit data (overhang and underhang) on the tibia for all templates will be taken from intra-operative measurements
Period: Overall Study
Arm/Group | iTotal CR TKR
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | iTotal CR TKR
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 32
Age, Continuous [Mean (Full Range); unit: Years] | 70.48 [57 to 87]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Women | 17

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Participants With a Customized Tibia Implant Displaying an Overhang of 3 mm or Greater
Description: Fit will be measured in 4 quadrants on the tibia using a ruler to measure the distance between the customized implant and the edge of the tibia.
Time Frame: Intraoperatively, up to 120 minutes
Population: 44 consecutive primary iTotal patients - number of patients with overhang of 3mm or more
Measure: Count of Participants; unit: Participants
Groups:
- Phase I: A series of 44 consecutive primary iTotal patients will be compared to assess the fit of the tibial tray intra-operatively. These patients will have a series of tibial templates from Standard TKR implant sets trialed on the operative knee. Each template will be optimally sized and positioned based on the surgeon's judgment. Implant fit data (overhang and underhang) on the tibia for all templates will be taken from intra-operative measurements
Arm/Group | Phase I
Number analyzed (Participants) | 44
Participants | 0

2. Primary Outcome: Phase II: Number of Participants With an Off-the-Shelf Implant Displaying an Overhang of 3 mm or Greater
Description: Fit will be measured in 3 quadrants on the tibia using a ruler to measure the distance between the off-the-shelf design and the edge of the tibia.
Time Frame: Intraoperatively, up to 120 minutes
Population: 44 consecutive primary iTotal patients - number of patients with overhang of 3mm or more
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled Subjects: A series of 44 consecutive primary iTotal patients will be compared to assess the fit of the tibial tray intra-operatively. These patients will have a series of tibial templates from Standard TKR implant sets trialed on the operative knee. Each template will be optimally sized and positioned based on the surgeon's judgment. Implant fit data (overhang and underhang) on the tibia for all templates will be taken from intra-operative measurements
Arm/Group | Enrolled Subjects
Number analyzed (Participants) | 44
Participants | 8

ADVERSE EVENTS:
Arm/Group | Enrolled Subjects
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No